CLINICAL TRIAL: NCT05686941
Title: Is Laryngeal Ultrasound a Useful Tool in the Assessment of Inducible Laryngeal Obstruction? A Protocol for a Two-stage Exploratory Pilot Study
Brief Title: Is Laryngeal Ultrasound Useful in the Assessment for ILO? A Protocol for a Two-stage Exploratory Pilot Study
Status: Recruiting | Type: Observational
Sponsor: Lancashire Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Edge Hill University (Other); University College, London (Other); Lancaster University (Other); University of Central Lancashire (Other)
Responsible Party: Principal Investigator, Claire Slinger, Consultant Speech & Language Therapist, Lancashire Teaching Hospitals NHS Foundation Trust
Other Study IDs: 298631
Record Dates: First submitted 2022-12-16; First posted 2023-01-17 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Vocal Cord Dysfunction; Asthma Brittle; Inducible Laryngeal Obstruction; Paradoxical Vocal Fold Motion
Keywords: Inducible laryngeal obstruction; Ultrasound
MeSH Terms: conditions — Vocal Cord Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Employees of the Host organisation in the Respiratory Team who meet the inclusion criteria
  Interventions: Other: Trans-cutaneous Laryngeal ultrasound (TLUS)
- Patients with suspected Inducible laryngeal Obstruction (ILO): Patients referred to a Tertiary referral centre who are suspected of having ILO
  Interventions: Other: Trans-cutaneous Laryngeal ultrasound (TLUS); Other: TLUS and simultaneous laryngoscopy

INTERVENTIONS:
Other: Trans-cutaneous Laryngeal ultrasound (TLUS) — Assessment of the larynx (specifically the vocal cords) with hand held portable ultrasound device to assess the movements of the vocal cords
Other: TLUS and simultaneous laryngoscopy — Assessment of the larynx (specifically the vocal cords) with hand held portable ultrasound device to assess the movements of the vocal cords with simultaneous video laryngoscopy (usual care)
  Other Names: TLUS
  Groups: Patients with suspected Inducible laryngeal Obstruction (ILO)

SUMMARY:
This study is a feasibility study to see if an ultrasound scan of the vocal cords can detect narrowing of the vocal cords as seen in a condition called inducible laryngeal Obstruction (the vocal cords narrow or close on breathing in, which makes it very difficult to breathe).

DETAILED DESCRIPTION:
This study aims to help understand whether viewing the vocal cords with an ultrasound device is useful to detect the movement of the vocal cords during breathing. This study is useful, as some people who have abnormal movements of the vocal cords on breathing in find it more difficult to breathe in, and often this leads to a big impact on their quality of life. It may also mean they are on medications that they may not need not be on, as abnormal movements of the vocal cords can often be mistaken for asthma, so they may have been placed on asthma medication when they may not need to be.

Usually, the way the abnormal movements of the vocal cords are seen now is via a small camera is placed via the nose into the throat to directly look at the vocal cords. Some people find this uncomfortable and may have to wait for a long time for it to happen. Also, this procedure is expensive, and is done in an endoscopy theatre, which may make it more daunting for some people, and make the wait longer. There are only a few centres that do these assessments with the camera, so people may have to travel some distance to have an assessment.

It is hoped, by doing this study, the investigators can see whether ultrasound can help assess if people have abnormal vocal cord movements when they breathe in. This will be done in 2 stages, one with healthy volunteers, and the second stage in patients who have been referred for assessment of their vocal cords to see if they have abnormal movements when breathing in. The investigators will also ask the volunteers and patients what their experience of having the ultrasound was like, and will ask the patients in the study how the ultrasound scan felt, when compared to the camera test

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* No definite signs or symptoms of vocal fold paralysis
* No voice change
* No history laryngeal surgeries
* No History of pathology
* No uncontrolled Respiratory disease

Exclusion Criteria:

* Participants with a known vocal fold pathology
* Participants with a history of head and neck surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * No definite signs or symptoms of vocal fold paralysis
  * No of history laryngeal surgeries
  * No history of pathology pathology
  * Too anxious to undergo procedure
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-06-27 (Estimated); Study Completion 2025-06-27 (Estimated)

PRIMARY OUTCOMES:
Number of vocal cords that are seen with the ultrasound | 1 day
  Can the vocal cord be seen under TLUS for Healthy Volunteers? Numeric data.
Number of particpants where visualisation of mimicked inspiratory adduction is visible on ultrasound | 1 day
  Can the vocal cords be seen to adduct under TLUS when healthy volunteers mimic ILO? Binary outcome: yes or no.
To assess the sensitivity, specificity and positive predictive value of the use of ultrasound | 1 day
  To assess the sensitivity, specificity and positive predictive value of the use of ultrasound in the assessment of ILO, using Laryngoscopy as reference standard in the patient population (n=30)
Questionnaire Investigating user perspectives on the acceptability of TLUS | 1 day
  A qualitative questionnaire investigating the patient and healthy volunteer perspectives on their experiences of undergoing TLUS assessment of the vocal cords. The questionnaire will look at the acceptability of the assessment in terms of comfort, repeatability, and comparison with laryngoscopy (for patients only).

CONTACTS AND LOCATIONS:
Overall Officials: Kina Bennett, Study Chair — Lancashire Teaching Hospitals NHS Trust; Claire Slinger, Principal Investigator — Lancashire Teaching Hospitals NHS Trust
Locations (1):
- Lancashire Teaching Hospitals NHS Trust, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT05686941/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT05686941/ICF_001.pdf